CLINICAL TRIAL: NCT03257189
Title: A Study to Evaluate the Performance, Usability, and Reliability of a Novel Device for Continuous Collection of Physiological Data in Healthcare and Remote Settings
Brief Title: Evaluation of Performance, Usability, and Reliability of a Novel Device for Continuous Collection of Physiological Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MC10 Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MC10-PTL-103
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Healthy Normals
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): This single arm consists of all subjects which will interact with the device under investigation as well as comparator devices.
  This includes the Physiological signal monitor intervention, Heart rate and heart rate variability comparison device intervention, Respiration rate comparison device intervention, and Activity classification intervention.
  Interventions: Device: Physiological signal monitor; Device: Heart rate and heart rate variability comparison device; Device: Respiration rate comparison device; Other: Activity classification

INTERVENTIONS:
Device: Physiological signal monitor — Wireless remote monitoring system intended for use by researchers and healthcare professionals for continuous collection of physiological data in home and healthcare settings.
Device: Heart rate and heart rate variability comparison device — FDA cleared reference device that monitors heart rate and heart rate variability in subjects
Device: Respiration rate comparison device — FDA cleared reference device that monitors respiration rate in subjects
Other: Activity classification — Visual annotation of subject posture and other activities used for reference

SUMMARY:
Study objective: The primary objective of the clinical investigation is to evaluate the accuracy of BioStamp nPoint system algorithm measurements.

Study design: A single-site, non-significant risk, open-label, prospective non-randomized clinical investigation designed to validate the accuracy of the various physiological parameters that the Wearable Sensor Patches acquire and the system processes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers, at least 18 years of age at the time of screening visit;
2. Fluent in English;
3. The subject is willing to comply with the protocol specified evaluations;
4. Subject is willing and cognitively able to sign informed consent

Exclusion Criteria:

1. Pregnancy;
2. Positive urine drug screen
3. History of active (clinically significant) skin disorders;
4. History of allergic response to silicones or adhesives;
5. Subjects with electronic implants of any kind (e.g. pacemaker)
6. History of sleep disorders or self-reported insomnia or other sleep conditions;
7. Broken, damaged or irritated skin or rashes near the sensor application sites;
8. Subjects that are MC10 employees or shareholders, or a spouse or child of an MC10 employee or shareholder;
9. Subjects who are physically or cognitively unable to normally perform activities of daily living, assessed at the discretion of the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTI Clinical Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via an established database at the clinical site, with the use of IRB approved flyers and posting on the clinical site website. The completely voluntary nature of participation in the study was emphasized.
  Subject recruitment and screening began July 17, 2017 and completed July 21, 2017.
Groups:
- Device Monitoring: This single arm consists of all subjects which will interact with the device under investigation as well as comparator devices.
  This includes the Physiological signal monitor intervention, Heart rate and heart rate variability comparison device intervention, Respiration rate comparison device intervention, and Activity classification intervention.
  Physiological signal monitor: Wireless remote monitoring system intended for use by researchers and healthcare professionals for continuous collection of physiological data in home and healthcare settings.
  Heart rate and heart rate variability comparison device: FDA cleared reference device that monitors heart rate and heart rate variability in subjects
  Respiration rate comparison device: FDA cleared reference device that monitors respiration rate in subjects
  Activity classification: Visual annotation of subject posture and other activities used for reference
Period: Overall Study
Arm/Group | Device Monitoring
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Subject sex documented at first visit to the clinic.
  Participants
    Female | 7
    Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Height (cm) [Mean (Standard Deviation); unit: centimeters] — Subject height measured and documented at first visit to the clinic.
  centimeters | 172.17 (8.61)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] — Subject weight measured and documented at first visit to the clinic.
  kilograms | 83.33 (11.63)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Subject BMI calculated from subject height and weight.
  kg/m^2 | 28.12 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Heart Rate Measured in Beats Per Minute Compared to Reference Device
Description: Heart rate as measured by the subject device in beats per minute will be compared to the reference device. The Mean Absolute Error (MAE) between measurements from each device is presented.
Time Frame: 2 days after informed consent
Population: Once comparator device malfunctioned resulting in a complete loss of Heart Rate data for one subject. All other subjects were analyzed, with n = 24 HR data pairs sampled at random (n = 8 samples each from sleeping, resting, and moving activities) per subject when available.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Device Monitoring
Number analyzed (Participants) | 29
beats per minute | 2.0 (5.1)

2. Primary Outcome: Accuracy of Heart Rate Variability Measured by Root Mean Square of Successive Differences (HRV RMSSD) Compared to the Reference Device
Description: Heart Rate Variability RMSSD is measured by the subject device determined by root mean square of successive differences in neighboring RR intervals and will be compared to the reference device. The Mean Absolute Error (MAE) between measurements from each device is presented.
Time Frame: 2 days after informed consent
Population: One comparator device malfunctioned, resulting in a complete loss of data for one subject. All other subjects were analyzed, with n = 24 HRV RMSSD data pairs sampled at random (n = 8 samples each from sleeping, resting, and moving activities) per subject when available.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Device Monitoring
Number analyzed (Participants) | 29
milliseconds | 5.1 (24.9)

3. Primary Outcome: Accuracy of Heart Rate Variability Measured by Low Frequency Content to High Frequency Content Ratio (HRV Ratio) Compared to the Reference Device
Description: HRV Ratio as measured by the subject device determined by low frequency content to high frequency content ratio (HRV Ratio) in beats per minute will be compared to the reference device. The Mean Absolute Error (MAE) between measurements from each device is presented.
Time Frame: 2 days after informed consent
Population: One comparator device malfunctioned, resulting in a complete loss of data for one subject. All other subjects were analyzed, with n = 24 HRV Ratio data pairs sampled at random (n = 8 samples each from sleeping, resting, and moving activities) per subject when available.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Device Monitoring
Number analyzed (Participants) | 29
unitless | 1.1 (1.8)

4. Primary Outcome: Accuracy of Respiration Rate Measured in Breaths Per Minute Compared to the Reference Device
Description: Respiration rate as measured by the subject device in breaths per minute will be compared to the reference device. The Mean Absolute Error (MAE) between measurements from each device is presented.
Time Frame: 2 days after informed consent
Population: All subjects were analyzed, with n = 8 total respiration rate data pairs sampled at random across the two nights of sleep per subject.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
breaths per minute | 1.3 (2.1)

5. Primary Outcome: Accuracy of Activity Classification as Compared to Visual Annotation
Description: The device under test will classify a subjects activity into sleeping, standing, sitting, lying, walking and other activities as the subject performs various predefined activities, which are annotated by an observer. The device's Activity Classification will be compared to the observer's annotation. The percentage of correct classifications by the device against indicated visual observation is presented. The percent correct is not a per subject average, but is the percentage of all activity classifications which were correct when compared to ground truth observation.
Time Frame: 2 days after informed consent
Population: All subjects were analyzed, with classifications compared against n = 5 clinician observed one minute long activities (lying, sitting, standing, walking, and stationary biking for "other" classification) per subject. For analysis of sleep classification accuracy, n = 5 one minute long samples were sampled across both nights of sleep per subject.
Measure: Number; unit: percent correct
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
percent correct | 98.7

6. Primary Outcome: Accuracy of Step Count Compared to an Observer's Manual Count
Description: The number of steps reported by the device under test during a 6 minute walk test will be compared to an observer's manual count of the number of steps taken.
Time Frame: 2 days after informed consent
Population: All subjects performed n=5 six minute walk tests on a treadmill. Instances in which the system classified the subject as "walking" for at least 95% of the activity were analyzed. The study device step count was compared to the manually observed step count, with the percent error of each test calculated. These errors were averaged and are presented.
Measure: Mean (Standard Deviation); unit: percent error
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
percent error | 2.4 (1.9)

7. Primary Outcome: Accuracy of Sleep Onset Time (Hours, Minutes, and Seconds), Sleep Wake Time (Hours, Minutes, and Seconds) as Compared to an Observer's Visual Annotation
Description: Sleep onset and wake times as reported by the device under test will be compared to an observer's visual annotation of the sleep onset and wake times. The Mean Absolute Error (MAE) between times as indicated by the device and observed times is presented.
Time Frame: 2 days after informed consent
Population: All subjects were analyzed, with n = 2 sleep onset and n = 2 sleep wake times compared per subject against sleep technician observations
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
minutes
  Sleep Onset | 6.8 (8.43)
  Sleep Wake | 11.5 (28.5)

8. Primary Outcome: Accuracy of Posture Classification as Compared to Visual Annotation
Description: The device under test will classify a subjects activity into sleep posture, standing posture, and sitting posture as the subject performs various predefined activities, which are annotated by an observer. The device's Posture Classification will be compared to the observer's annotation. The percentage of correct classifications by the device against indicated visual observation is presented. The percent correct is not a per subject average, but is the percentage of all posture classifications which were correct when compared to ground truth observation.
Time Frame: 2 days after informed consent
Population: All subjects were analyzed, with each subject completing n = 5 repetitions of each sleeping / lying (supine, prone, lying left, lying right) and sitting / standing (upright, leaning backward, leaning forward, leaning left, leaning right) postures.
Measure: Number; unit: percent correct
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
percent correct | 92.9

9. Primary Outcome: Number of Sensors That Remained Sufficiently Adhered to Subjects for 24 Hours as Assessed by a 5 Point Scale
Description: The level of sensor adhesion will be assessed by a 5 point scale (0- sensor is greater than or equal to 90% of sensor adhered, 4-sensor completely detached from subject). Sensors receiving scores of 0 and 1 will be determined to have acceptable adhesion, while scores of 2, 3, and 4 will be considered unacceptable adhesion. The percentage of sensors which had acceptable adhesion at sensor removal is presented.
Time Frame: 2 days after informed consent
Population: All subjects analyzed, with 6 sensor locations per subject evaluated for adhesion to skin at device removal. Subjects wore n = 4 sensors (two sensors at chest and thigh locations required for algorithmic outputs, and one sensor at shank and one at forearm locations) on Day 1 and n = 2 sensors (chest and thigh algorithm location sensors) on Day 2.
Measure: Number; unit: percent passing
Units Other Than Participants: Total Sensors Evaluated for Adhesion
Arm/Group | Device Monitoring
Number analyzed (Participants) | 30
Number analyzed (Total Sensors Evaluated for Adhesion) | 180
percent passing
  All Sensors | 83
  Sensors for Algorithm Outputs (Chest and Thigh) | 92

ADVERSE EVENTS:
Time Frame: Adverse event data was available for collection for 3 days after the subject left the clinic. Subjects were evaluated throughout their 3 days at the clinic and a safety follow up phone call was conducted 3 days after their last clinic visit.
Description: All adverse events (all-cause mortality, serious, and non-serious) were collected. The study was inherently low risk, as the test device is a non-significant risk device and study population was limited to healthy volunteers.
Arm/Group | Device Monitoring
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Monitoring (N=30)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A single non-serious adverse event was reported during the evaluation period. A subject self reported mild nasal congestion after spending the night at the clinical site. This was deemed unrelated to the test device.

LIMITATIONS AND CAVEATS:
This study design was based off of the predicate device's pivotal study design. It was limited to healthy subjects only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03257189/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03257189/SAP_001.pdf